CLINICAL TRIAL: NCT06565936
Title: Clinical Application of DPA-714 and FDG PET/MRI Imaging in Patients With Depression
Brief Title: DPA-714 and FDG PET/MRI in Depression
Acronym: DAF-PMID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PJ-KS-KY-2024-153(X)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Magnetic Resonance Spectroscopy; Product Labeling; N,N-diethyl-2-(2-(4-(2-fluoroethoxy)phenyl)-5,7-dimethylpyrazolo(1,5-a)pyrimidin-3-yl)acetamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recurrent depression patients group (Experimental): Evaluation of neuroinflammation and cerebral metabolism in the prefrontal cortex, anterior cingulate cortex, insula, and other brain regions of interest in patients with recurrent depression.
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714 or [18F]F-FDG
- First-episode depression patients group (Experimental): Evaluation of neuroinflammation and cerebral metabolism in the prefrontal cortex, anterior cingulate cortex, insula, and other brain regions of interest in patients with first episode depression.
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714 or [18F]F-FDG
- Healthy controls group (Other): Evaluation of neuroinflammation and cerebral metabolism in the prefrontal cortex, anterior cingulate cortex, insula, and other brain regions of interest in healthy controls.
  Interventions: Radiation: PET scan with tracer injection [18F] DPA-714 or [18F]F-FDG

INTERVENTIONS:
Radiation: PET scan with tracer injection [18F] DPA-714 or [18F]F-FDG — Brain PET/MRI imaging will be conducted following the administration of [18F] DPA-714 or [18F]F-FDG. The radiopharmaceuticals are given intravenously in doses that are safe for the human body, with minimal quantities to reduce potential effects. Additionally, the irradiation levels are kept low, ensuring the procedure is safe and reliable for patients.

SUMMARY:
Depression, a common psychological disorder, is characterized by persistent low mood, loss of interest, and anhedonia, leading to significant dysfunctions and a high suicide risk. Its pathogenesis remains challenging, with recent focus on neuroinflammation-a chronic immune response in the central nervous system-as a potential contributor. PET imaging, using tracers like 18F-FDG and [18F]DPA-714, can visualize metabolic and neuroinflammatory changes. Combining these two tracers can explore the correlation between neuroinflammation and glucose metabolism in depression, further elucidating its possible mechanisms. We hypothesize that microglial activation in depression, especially in major gray matter regions of interest (prefrontal cortex, anterior cingulate cortex, and insula) and 12 additional regions and subregions, will show higher TSPO levels and increased glucose metabolism compared to the control group.

DETAILED DESCRIPTION:
Depression is a common psychological disorder caused by various factors, characterized by significant and persistent low mood, loss of interest, and anhedonia as core symptoms, leading to physical, psychological, and social dysfunctions, with a high risk of suicide. The pathogenesis of depression remains a challenging topic in the medical field. Imaging studies are crucial for exploring the pathogenesis of depression. Recently, neuroinflammation has gained significant attention regarding the pathophysiological mechanisms of depression. Neuroinflammation, a chronic inflammatory response of the immune system in the central nervous system, may be related to the onset and progression of depression. PET is an imaging method that uses radioactive tracers to visualize physiological activities and metabolic processes in the body. 18F-FDG-PET can reflect neuronal degeneration and the reduction in the number and function of protrusions in vitro, directly indicating lesion sites and involvement. Therefore, PET/MRI brain metabolism imaging can uncover possible pathogenesis and explore unique brain network characteristics from a molecular imaging perspective. PET studies can depict local functional metabolism and neurochemical changes in the brain through radionuclide labeling. [18F]DPA-714, a PET tracer, is a high-affinity ligand for the translocator protein (TSPO), a mitochondrial outer membrane protein expressed in activated microglia and macrophages in the brain, serving as a marker of neuroinflammation. As a TSPO radioligand, DPA-714 can explore in vivo changes in neuroinflammation. Combining these two tracers can explore the correlation between neuroinflammation and glucose metabolism in depression, further elucidating its possible mechanisms.

This study will collect data from patients diagnosed with recurrent depression and first-episode depression in the Psychosomatic Sleep Department and Neurology Department of the First Affiliated Hospital of Dalian Medical University. Healthy individuals who underwent "DPA-714 or FDG imaging PET/MRI" physical examinations in the PET/CT room of our hospital will also be included. According to the inclusion and exclusion criteria, the groups will consist of 25 cases of recurrent depression, 25 cases of first-episode depression, and 20 healthy controls. Additionally, all three groups will undergo neuropsychological assessments, including Hamilton Anxiety Scale, Hamilton Depression Scale, Mini-mental State Examination, Montreal Cognitive Assessment, Pittsburgh Sleep Quality Index Scale, and other related cognitive, sleep, and emotional scales. We used DPA-714 imaging agent PET/MRI to scan the whole brain, selecting major gray matter regions of interest (prefrontal cortex, anterior cingulate cortex, and insula) and 12 additional regions and subregions to measure TSPO values. The patients with recurrent depression and first episode depression were compared with the normal control group to explore their characteristics. Moreover, through the relationship between TSPO values and neuropsychological scores, the correlation between TSPO values and depression severity was explored.

The statistical method we use is that SPSS26.0 statistical software (IBM, New York, United States) was used to conduct statistical analysis on the basic demographic data of each group. Normal test and homogeneity test of variance were performed on the data. Continuous variables conforming to normal distribution were expressed in the form of mean ± standard deviation (±s). Samples that do not conform to a normal distribution and variables represented as graded data are described by the median (interquartile range). The Chi-square test was used to compare categorical data groups. For normally distributed data, a two independent sample T-test was employed. Non-normally distributed data were analyzed using the Mann-Whitney U test. Pearson or Spearman correlation coefficients were used for correlation analysis, depending on the data distribution.

ELIGIBILITY:
Inclusion Criteria:

1. For all groups :

   * No alcohol or psychoactive substances such as coffee had been consumed in the 24 hours prior to the examination
   * MMSE≥24 points，MOCA≥26 points
   * No anti-infective drugs in the past 1 month, no cold, fever or other infection history in the past 2 weeks
   * Patients with diabetes had fasting controlled below 9.0mmol/L before the examination
   * Volunteer to participate in the study and sign the informed consent
2. For Recurrent depression patients:

   * Meet the Diagnostic criteria for recurrent major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
   * Age 35-85 years old, gender is not limited
   * HAMD≥8 points
3. For first episode depression Patients:

   * Gender, age and education level were matched with the recurrent depression group
   * Meet the Diagnostic criteria for the first episode of depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
   * HAMD≥8 points
4. For controls:

   * Healthy people undergoing "DPA-714 or FDG imaging PET/MRI" physical examination in PET/CT room of our hospital
   * Gender and education level were consistent with both the recurrent depression group and the first-episode depression group
   * never used any psychotropic drugs
   * HAMD<8 points；HAMA<7 points

Exclusion Criteria(for all groups):

* Have a history of organic mental disorders or other mental disorders
* A family history of hereditary diseases
* Persons with mental retardation or dementia
* A history of psychoactive substance abuse
* Can not cooperate with/complete the psychological examination scale
* Previously found serious physical diseases (heart, brain, liver, lung and kidney)
* MRI contraindications, abnormalities found in head CT or MRI
* A history of drug or alcohol abuse
* Have a history of metabolic diseases such as hyperthyroidism, hypothyroidism,and rheumatic diseases
* are in the state of pregnancy or breastfeeding

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of baseline and follow up regional brain TSPO levels and cerebral metabolism using PET/MRI | for 2 years
  TSPO values for the major gray matter regions of interest (prefrontal cortex, anterior cingulate cortex, and insula) and 12 additional regions and subregions were observed in patients with recurrent and first-episode depression compared to controls.Estimates of brain TSPO concentrations measured with PET will serve as a marker for neuroinflammation. Variation of the regional cerebral glucose consumption and TSPO-PET measures will be compared between three groups.

SECONDARY OUTCOMES:
Mini-Mental State Evaluation (MMSE) | for 2 years
  Clinician-administered screening tool used to systematically and thoroughly assess mental status through five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Scores range between 0-30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Scores of Hamilton Depression Scale | for 2 years
  Using to assess depressive symptoms. With higher scores associated with more severe depression symptoms. Total scores <8 is normal; Mild depression with total scores of 8～17; Moderate depression with total scores of 18～24; Total scores >24 for severe depression.
Scores of Hamilton Anxiety Scale | for 2 years
  Using to assess anxiety symptoms. With higher scores associated with more severe anxiety symptoms. Total scores< 7 indicates no anxiety; Total scores≥7 indicates possible anxiety; Total scores≥14 indicates anxiety; Total scores≥21 indicates obvious anxiety; Total scores≥29 points indicates serious anxiety.
Pittsburgh Sleep Quality Index | for 2 years
  Using to assess the sleep quality. Total scores of 0-5 indicates that the quality of sleep is very good, 6～10 indicates that the quality of sleep is OK, 11～15 indicates that the quality of sleep is average, and 16～21 indicates that the quality of sleep is poor.
Correlation between microglial activation and cerebral metabolism in the prefrontal cortex, anterior cingulate cortex, insula, and other regions of interest, and the severity of disease in patients. | for 2 years
  Patients will be followed up longitudinally to monitor changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Zhang, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No